CLINICAL TRIAL: NCT03528447
Title: The Effect of Pulmonary Rehabilitation on Cognitive Status in Lung Transplantation Candidates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR_cognition
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment; Pulmonary Rehabilitation
Keywords: lung transplantation; cognition; MOCA; exercise; pulmonary rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Lung transplantation candidates who refered from Lung Transplantation surgery team will undergo the Pulmonary Rehabilitation program for 3-months (2 days at hospital, 3 days at home). Patient will evaluate at the beginning and end of the program.Cognitive functions and exercise capacities of the patients before and after the program will be evaluated.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Aerobic training:The aerobic exercise program consists of treadmill walking, cycle ergometer and arm ergometer training. Group exercises were performed in sets of 15 minutes each with three exercise modalities.
  Strength training:It is recommended that resistance targets are set at loads equivalent to 20 to 40% of a 1-repetition maximum (1RM) maneuver and performed between 8 to 12 repetitions for 1 to 2 sets per session.
  Home exercise programme:The program included breathing exercises (local expansion exercises, diaphragmatic breathing and pursed lip breathing), free walking, upper and lower extremity strengthening exercises with Thera-Band.

SUMMARY:
Pulmonary rehabilitation program with aerobic and strengthening for 3 months will be applied to the candidates for lung transplantation. The program will be designed to be 2 days supervised weekly and 3 day home program. Cognitive functions and exercise capacities of the patients before and after the program will be evaluated.

DETAILED DESCRIPTION:
The fact that cognition is not always included in the assessment routine makes it difficult to clarify which patient group or severity of illness is more affected by this issue. The effect of exercise on cognitive functions is a remarkable issue in recent years. It can also be predicted that cognitive function may be effective on program adaptation in patients who are given home program without supervision. The aim of the investigator's study was to investigate the effect of pulmonary rehabilitation on cognitive status in candidate lung transplant recipients.

Lung transplantation candidates who refered from Lung Transplantation surgery team will receive the Pulmonary Rehabilitation program for 3-months (2 days at hospital, 3 days at home). Exercise program includes aerobic (walking band, bicycle, arm ergometer) and strengthening (with free weights) components. Patient will evaluate at the beginning and end of the program. Demographic information, diagnosis distributions, educational status of patients will be recorded. Exercise capacities are determined by 6 min walk test. The medical research concil dyspnea scale is used in determining the dispense levels. Montreal Cognitive Function Assessment (MOCA) is used to determine cognitive functions. Cognitive functions and exercise capacities of the patients before and after the program will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To be listed for lung transplantation,
* Pulmonary rehabilitation exercise program planned to be taken,
* Volunteers who have agreed to participate in the work,
* Patients who can complete the 3-month Pulmonary Rehabilitation program.

Exclusion Criteria:

* Failure to complete the planned exercise program for any reason,
* Not to be literate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline distance covered in six minute walking test at 3-months. | 6 minute
Change from baseline The Montreal Cognitive Assessment (MoCA) at 3-months | 15 minute
  The Montreal Cognitive Assessment (MoCA; Nasreddine et al., 2005) takes approximately 10 minutes to administer and was designed to detect mild cognitive impairment.Thirty items assessing multiple cognitive domains are contained in the MoCA: short-term memory (5 points); visuospatial abilities via clock drawing (3 points), and a cube copy task (1 point); executive functioning via an adaptation of Trail Making Test Part B (1 point), phonemic fluency (1 point), and verbal abstraction (2 points); attention, concentration, and working memory via target detection (1 point), serial subtraction (3 points), digits forward (1 point), and digits backward (1 point); language via confrontation naming with low-familiarity animals (3 points), and repetition of complex sentences (2 points); and orientation to time and place (6 points) (Nasreddine et al., 2005). The MoCA is scored by obtaining an item total and the authors recommend a clinical cutoff score of 26.

SECONDARY OUTCOMES:
Change from baseline modified Medical Council Dyspnea score at 3-months | 5 minute
  The scale will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 3-months | 20 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)